CLINICAL TRIAL: NCT02552394
Title: Anti-Prostate-Specific Membrane Antigen Monoclonal Antibody J591 in Patients With Advanced Prostate Cancer and Unfavorable Circulating Tumor Cell Counts
Brief Title: J591 in Patients With Advanced Prostate Cancer and Unfavorable Circulating Tumor Cell Counts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1503015998
Record Dates: First submitted 2015-08-03; First posted 2015-09-17 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — J591 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HuJ591 Administration (Experimental): 6 subjects will be treated at 300 mg dose. The decision about treating subjects at the lower dose will depend upon their response. If ≥4 of 6 subjects respond at the 300 mg level, then 6 more subjects will be recruited at the 200 mg level. If ≥4 of 6 subjects respond at the 200 mg level than 6 more subjects will be recruited at the next dose level of 100 mg. If ≥ 4/6 subjects respond at this level, then 6 subjects will be recruited at the last dose level of 50 mg. At any level, if the first four consecutive subjects respond, the next two subjects will be enrolled in the same dose-level cohort and further subjects will be recruited at the next dose level. Response at every dose level is defined by conversion from an unfavorable CTC count at baseline to a favorable CTC count.
  Interventions: Drug: huJ591

INTERVENTIONS:
Drug: huJ591 — HuJ591 will be administered as an intravenous infusion at a concentration of 5 mg/mL and rate of <5 mg/minute. Pre-medications prior to J591 infusion with diphenhydramine 25 - 50 mg p.o. or IV and acetaminophen 500 - 650 mg p.o.
  Other Names: J591

SUMMARY:
This clinical trial is for men with advanced prostate cancer that may have spread to other parts of the body.

Currently, once prostate cancer cells have spread from the prostate to other organs it is not treatable by surgery. The purpose of this study is to treat patients with an experimental antibody (i.e. that has not been FDA approved) called J591 that attaches itself to a special protein on cancer cells called PSMA to try to eliminate these cancer cells (called circulating tumor cells) from the circulation.

In the initial phase of the study, 6 participants will receive the experimental J591 treatment. Routine blood tests, research blood tests, physical exam will be performed at each visit. Participants will also be asked to complete a questionnaire about how they are feeling. Participants will have a radiographic scan every 3 months to check the status of their disease.

Participants who tolerate the treatment well may be re-treated at the same level every 3 months, and may continue on treatment as long as they are responding to therapy and not experiencing unacceptable side effects.

DETAILED DESCRIPTION:
J591 is a de-immunized monoclonal antibody against the extracellular domain of prostate-specific membrane antigen (PSMA). Background data demonstrate that mAb Hu-J591 doses as low as 20 mg may lead to a decrease in CTCs and that doses up to 300 mg are safe. With a goal of establishing less frequent, potentially more convenient and cost-effective future therapy, the investigators propose a single-center, open-label, dose de-escalation study to determine the effect of mAb Hu-J591 on circulating tumor cells in subjects with metastatic PC. Four dose levels are planned with a minimum of 6 and maximum of 24 subject enrollment starting with a single infusion of 300 mg of mAb Hu-J591.

In the initial phase of the study a cohort of 6 subjects will receive 300 mg of mAb Hu-J591 and blood samples will be collected pre and post-infusion for the detection of CTCs, PSA and to assess hematological toxicity at screening, baseline, week 1, week 4, week 8, and week 12. In addition, patients will receive a dose of 89Zr-DFO-huJ591 (5 mCi) 2-4 weeks prior to treatment and will undergo 89Zr-DFO-huJ591 PET imaging 1-3 weeks pre-treatment (optional) as well as repeat 89Zr-DFO-huJ591 infusion (5 mCi) at 11 weeks and PET/CT imaging at 12 weeks (optional).

If less than four subjects respond by dropping their CTC counts from more than or equal to 5 CTCs/7.5 mL whole blood to less than 5 CTCs/7.5 mL whole blood in the initial cohort, the trial will be ended at this dose. If four or more subjects respond, an additional 6 subjects will be accrued to the second dose level (200 mg). The same decision rule will be applied to evaluate two additional lower dose levels (100 mg, 50 mg) with 6 subjects enrolled in each cohort. Imaging studies will be performed prior to treatment at screening and at 3 months or as clinically indicated to assess disease response.

Subjects who tolerate the initial infusion well (< grade 2 toxicities) may be re-treated every 3 months (12 weeks) at the same dose-level until progression.

ELIGIBILITY:
Inclusion Criteria

1. Histologic/Cytologic diagnosis of prostate carcinoma
2. Subject must have progressive metastatic prostate cancer as defined as at least any one of the following:

   * New lesions on bone scan
   * Progression of disease on CT/MRI as defined by RECIST
   * PSA progression defined by an absolute value 2 ng/mL with an increase in PSA determined by two separate measurements taken at least one week apart and confirmed by a third, and if necessary, a fourth measurement. If the third measurement is not greater than the second measurement, then a fourth measurement must be taken; the fourth measurement must be greater than the second measurement for the subject to be eligible for enrollment in the study. Furthermore, the confirmatory PSA measurement (i.e., the third or, if applicable, fourth PSA measurement) must be 2 ng/mL and ≥ 25% above the previous nadir.
   * Increase in circulating tumor cell (CTC) count via CellSearch methodology in the absence of responding tumor by other criteria.
3. Subjects must remain on a stable hormonal therapy regimen.

   * Subjects who have received traditional anti-androgen (i.e. bicalutamide, nilutamide, flutamide) therapy with a resulting PSA decline must continue anti-androgen therapy or demonstrate progression following discontinuation of anti-androgen therapy (not necessary for those who never responded to anti-androgen addition).
   * Medical or surgical castration will be continued for the duration of the trial in all subjects.
   * Subjects who have any measure of progression on androgen receptor signaling inhibitors (such as enzalutamide or apalutamide) or CYP17 inhibitors (such as abiraterone acetate) and wish to continue must remain on a stable regimen.
4. CTCs ≥ 5 per 7.5ml of whole blood performed by CellSearch system within 1 month of enrollment (may be performed as part of screening).
5. Subjects capable of fathering children must agree to use an effective method of contraception for the duration of the trial.

Exclusion Criteria

1. Prior cytotoxic chemotherapy and/or radiation therapy within 4 weeks of treatment
2. AST or ALT > 2.5x ULN unless secondary to liver metastasis (then AST/ALT > 5x ULN is exclusionary provided subject meets bilirubin requirements)
3. Bilirubin (total) > 1.5x ULN; subjects with known Gilbert's syndrome are eligible if direct bilirubin is within normal limits
4. Serum Creatinine > 3x ULN
5. Absolute Neutrophil Count <1000/µL
6. Hemoglobin <8 g/dL
7. Platelet Count <50,000/µL
8. ECOG Performance Status >2
9. Life expectancy < 6 months
10. Any serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which in the investigator's opinion might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
11. Prior investigational therapy (medications or devices) within 4 weeks of treatment. Furthermore, other investigational anti-cancer therapy is not permitted during the treatment phase.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Changes in frequency of achieving a decrease in Circulating tumor count (CTC) | CTCs will be measured on Day 1, Day 8, Day 29, Day 57, and Day 85, then monthly until the date of first documented progression, or death from any cause, whichever came first assessed up to 100 months
  Determine the effect of mAb Hu-J591 on reducing circulating tumor cells (CTCs) from > 5/7.5 mL of whole blood to < 5/7.5 mL of whole blood in metastatic prostate cancer (PC) with elevated baseline CTC count and to identify the least effective dose that clears CTCs.

SECONDARY OUTCOMES:
Changes in prostate specific antigen (PSA) measurable disease response | Response will be measured by performing CT scans every 3 months from baseline until the date of first documented progression, or death from any cause, whichever came first assessed up to 100 months
  Dose cohort will report the proportion of subjects achieving declines of ≥ 30% confirmed by a second PSA value ≥ 2 weeks later. In addition, for subjects with measureable disease at baseline, the frequency of achieving an objective response as described by Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) will be presented by dose cohort. The distributions of the duration of both of these clinical outcomes will be presented by dose level.
Change in duration of Circulating tumor count (CTC) response | Labs will be collected at Screening, Day 1, Day 8, Day 29, Day 57 and Day 85
  Descriptive statistics (e.g. means, proportions, medians, range) will be calculated to summarize the baseline CTC values and the change at 12 weeks and presented by dose level. This will include calculating the frequency of CTC responders, the proportion of responders, the percent change in CTC count, the duration of CTC count remaining <5/7.5mL if it occurs, the duration of time to first measurement of CTC count <5/7.5mL.
Change in disease response through the optional (but recommended) prostate specific membrane antigen (PSMA) PET/CT imaging | Performed prior to treatment at screening and at 3 months/12 weeks or as clinically indicated
  Measurable disease response will be calculated using Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) with Prostate Cancer Clinical Trials Working Group 3 (PCWG3) modifications.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No